CLINICAL TRIAL: NCT06402721
Title: An Open-label Study to Evaluate the Pharmacokinetics, Safety and Tolerability of BAY 3283142 in Participants With Impaired Hepatic Function (Classified as Child-Pugh A or B) in Comparison to Matched Controls With Normal Hepatic Function
Brief Title: A Study to Learn About How BAY 3283142 Moves Into, Through, and Out of the Body After a Single Dose in Participants With Reduced Liver Function Compared to Participants With Normal Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22129
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Disease; Hepatic Impairment
Keywords: CKD
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Mild hepatic impairment (Experimental): Participants with mild hepatic impairment.
  Interventions: Drug: BAY3283142
- Group 2: Moderate hepatic impairment (Experimental): Participants with moderate hepatic impairment.
  Interventions: Drug: BAY3283142
- Group 3 and 4: Normal hepatic function (control group) (Experimental): Control group(s) of age-, weight-, and gender-matched participants with normal hepatic function.
  Interventions: Drug: BAY3283142

INTERVENTIONS:
Drug: BAY3283142 — Single oral dose.

SUMMARY:
Researchers are looking for a better way to treat people who have chronic kidney disease (CKD).

CKD is a condition in which the kidneys' ability to work properly gradually decreases over time. The kidneys help the body get rid of waste through urine and filter the blood before sending it back to the heart. When kidney function decreases, waste builds up in the body, which can cause various complications.

The study treatment, BAY 3283142, is under development to treat CKD. It works by activating a protein called soluble guanylate cyclase (sGC) that generates cGMP - a molecule that relaxes blood vessels and is thought to have beneficial effects in CKD. BAY3283142 is broken down in the liver by a specific enzyme before it is removed from the body.

In this study, researchers want to understand how a mild or moderate reduction in liver function affects the blood levels of BAY3283142.

The main purpose of this study is to learn how BAY3283142 moves into, through, and out of the body, after a single dose of BAY3283142 in participants with reduced liver function.

For this, the researchers will analyze:

* Area under the curve (AUC): a measure of the total amount of BAY3283142 in participants' blood over time
* Maximum observed concentration (Cmax): the highest amount of BAY 3283142 in participants' blood The AUC and Cmax values for participants with reduced liver function will be compared with the values for participants with normal liver function.

The study participants will be assigned to one of the four treatment groups based on their liver function:

* Group 1: participants with mild reduction in liver function
* Group 2: participants with moderate reduction in liver function
* Groups 3 and 4: participants with normal liver function who will be matched for age, weight, and gender with participants with reduced liver function All participants will take a single dose of BAY3283142 as a tablet by mouth without food.

Each participant will be in the study for around 5 to 6 weeks, which includes:

* a visit within 28 days of starting treatment to confirm if the participant can take part in this study
* a hospital stay for 7 days during which the participant will be given a single dose of BAY3283142 and the study doctor will monitor the participant's health
* a visit after 7 to 10 days of taking BAY3283142 during which the study doctor will perform a health check-up on the participant

During the study, the doctors and their study team will:

* check participants' health by performing tests such as blood and urine tests, blood pressure measurements, and checking heart health using an electrocardiogram (ECG)
* ask the participants questions about how they are feeling and what adverse events they are having An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events, irrespective of whether they think it is related or not to the study treatment.

Access to study treatment after the end of this study is not planned. Participants with liver problems can continue taking their other prescribed medicines as usual.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 79 years (both inclusive) at the screening visit
* Participants with hepatic impairment classified as Child-Pugh A or B

  * Disease confirmed by histopathology, (e.g. previous liver biopsy), laparoscopy, CT, MRI, ultrasound or fibroscan
  * Stable liver disease in the last 2 months
* Participants who have normal hepatic function and are overtly healthy.
* Body mass index (BMI): 18 to 36 kg/m*2 (both inclusive).
* Male or female. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

  * Male participants: Must agree to use contraception/barrier as detailed below:

    * Agree to use a male condom and should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak when having sexual intercourse with a woman of childbearing potential who is not currently pregnant.
    * Agree to use a male condom when engaging in any activity that allows for passage of ejaculate to another person.
  * Female participants: A female participant is eligible to participate if she is not pregnant or breast feeding, and one of the following conditions applies:

    * Is a woman of nonchildbearing potential (WONCBP)
    * Is a women of childbearing potential (WOCBP) and using a contraceptive method that is highly effective (with a failure rate < 1% per year), with low user dependency, starting from signing the informed consent form and for at least 10 days after the intake of study intervention. The investigator should evaluate the potential for contraceptive method failure (e.g. noncompliance, recently initiated) in relationship to the dose of study intervention.
* A WOCBP must have a negative highly sensitive pregnancy test within 24h before the first dose of study intervention.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

* Severe ascites of more than 6 L (estimated by ultrasound)
* Evidence of hepatic encephalopathy related to chronic liver disease > grade 2 (exclusion by Number Connection Test).
* Renal failure with an estimated glomerular filtration rate ≤40 mL/min (according to CKD-EPI equation).
* Relevant diseases within the last 4 weeks prior to first study drug intervention.
* Acute diarrhea or constipation within 14 days before the predicted first dosing day.
* Febrile illness within 2 weeks prior to the admission of the study center
* Tendency for vasovagal reactions (e.g. after venipuncture) or syncope.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-05-17 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of BAY3283142 | On Day 1 (dosing day), Day 2, Day 3, Day 4, Day 5, and Day 6.
  AUC(0-tlast) will be used as main parameter, if mean AUC cannot be reliably determined in all participants.
Maximum observed drug concentration (Cmax) of BAY3283142 | On Day 1 (dosing day), Day 2, Day 3, Day 4, Day 5, and Day 6.

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events | 7 days after last administration of study drug

CONTACTS AND LOCATIONS:
Locations (1):
- Orlando Clinical Research Center (OCRC), Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.